CLINICAL TRIAL: NCT04058886
Title: Easing the Burden of Dementia Caregiving: A Telephone-delivered Mindfulness Intervention for Rural, African American Families
Brief Title: Telephone-delivered Mindfulness Intervention for African American Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-0053; R21AG061728 (NIH)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Dementia; Caregiver; Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telephone-delivered Mindfulness (Experimental): Participating caregivers and care partners will receive mindfulness training in 8 weekly telephone sessions plus one retreat. Respite care for the care recipient is provided for the retreat.
  Interventions: Behavioral: Telephone-delivered Mindfulness

INTERVENTIONS:
Behavioral: Telephone-delivered Mindfulness — The telephone-delivered mindfulness training intervention that will incorporate the following elements: 1) training for primary caregivers (CG) and their caregiving partner (CP) in a telephone-based mindfulness training intervention; 2) groups of up to eight participants (four CG-CP pairs) plus an instructor, on a shared telephone line; and 3) training in a 8-week, modified MBSR program, which places additional emphasis on training in the following: a) mindful experiencing, including mindfulness of feelings and body sensations; b) mindful communication, including non-verbal mindfulness, mindful listening, and mindful speaking; and c) mindful compassion for self and others. Additionally, homework assignments will involve listening to exercises on a dial-in telephone line; and assignments for CG-CP dyads (e.g. mindful listening and communication practices) as well as CG mindfulness practices in the presence of care recipients (e.g. mindful eating, and mindful listening).

SUMMARY:
This study is assesses the feasibility and acceptability of telephone-delivered mindfulness training designed to alleviate caregiver burden for African-American rural caregivers of individuals with moderate to severe dementia, as defined by the caregiver. The study utilizes a single-group, uncontrolled design to test the feasibility and acceptability of the intervention for the target population.

DETAILED DESCRIPTION:
Mindfulness interventions can decrease caregiver burden and improve coping skills, including decreased emotion-based coping, increased tolerance for uncertainty, improved psychological well-being and quality of life while potentially improving relationship quality and communication.

This study utilizes a single-group, uncontrolled design to assess the feasibility and acceptability of telephone-delivered mindfulness training designed to alleviate caregiver burden for African-American rural caregivers of individuals with moderate to severe dementia, as defined by the caregiver. The telephone-delivered mindfulness intervention will improve geographical access for rural caregivers and deem more flexible for a caregiver's schedule. The study's intervention consists of mindfulness training delivered by telephone once weekly for 8 weeks. The intervention also includes one retreat for which respite care will be provided, if needed. The intervention, based on, Kabat-Zinn's mindfulness-based stress reduction (MBSR), will emphasize the following: 1) mindful experiencing, including mindfulness of feelings and body sensations; 2) mindful communication, including non-verbal mindfulness, mindful listening, and mindful speaking; and 3) mindful compassion for self and others.

ELIGIBILITY:
Inclusion Criteria:

* The candidate is at least 18 years old;
* The candidate self-identifies as Black or African American;
* The candidate provides at least 4 hours of care per day to the care recipient, who must have either a diagnosis of dementia OR have a score of at least 2 or higher on the Alzheimer's Disease Screening tool (AD-8) or a score of 8 or higher on the Functional Assessment Staging of Alzheimer's disease (FAST) scale (indicative of moderate - severe dementia);
* The candidate is able to identify and recruit an additional informal caregiver (care partner) to participate in the study. The care partner must consider themselves as part of the caregiving team that helps to make decisions about the care of the care recipient. The care partner may be a blood relative or close friend, but not a formal caregiver. The care partner need not live in the same geographic area.
* Both the candidate primary caregiver and care partner must have access to a telephone and express a willingness to participate in the pre- and post-participation assessments, the intervention calls, and the intervention retreat.

Exclusion Criteria:

* The candidate is too unwell to participate; e.g., with an active diagnosis of cancer or more than 3 hospitalizations in the past year;
* The primary caregiver is unable to identify and recruit a care partner willing to commit to the study requirements;
* The care recipient does not meet the criteria for dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gaylord, PhD, Principal Investigator — UNC-Chapel Hill; Sharon Williams, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Program on Integrative Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Faurot KR, Roth I, Harr E, Shafer J, Giscombe K, Sheffield-Abdullah KM, Lathren C, Brantley M, Williams SW, Gaylord SA. Feasibility of a Telephone-Delivered Mindfulness Intervention for Informal Caregivers of Rural-Dwelling African Americans With Dementia. Glob Adv Integr Med Health. 2025 Jun 4;14:27536130251347944. doi: 10.1177/27536130251347944. eCollection 2025 Jan-Dec. PMID 40475373

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary Caregivers and Care Partners were enrolled as dyads. A total of 28 dyads and 1 additional Primary Caregiver were included in the analysis. One Care Partner was not enrolled as planned after the Primary Caregiver had already been enrolled.
Groups:
- Telephone-delivered Mindfulness: Participating caregivers and care partners will receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
  Telephone-delivered Mindfulness: The telephone-delivered mindfulness training intervention that will incorporate the following elements: 1) training for primary caregivers (CG) and their caregiving partner (CP) in a telephone-based mindfulness training intervention; 2) groups of up to eight participants (four CG-CP pairs) plus an instructor, on a shared telephone line; and 3) training in a 8-week, modified Mindfulness-Based Stress Reduction (MBSR) program, which places additional emphasis on training in the following: a) mindful experiencing, including mindfulness of feelings and body sensations; b) mindful communication, including non-verbal mindfulness, mindful listening, and mindful speaking; and c) mindful compassion for self and others. Additionally, homework assignments will involve listening to exercises on a dial-in telephone line; and assignments for CG-CP dyads (e.g. mindful listening and communication practices) as well as CG mindfulness practices in the presence of care recipients (e.g., mindful eating, and mindful listening).
Period: Overall Study
Arm/Group | Telephone-delivered Mindfulness
Started | 57
Primary Caregivers Started | 29
Care Partners Started | 28
Primary Caregivers Completed | 27
Care Partners Completed | 25
Completed | 52
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Inadequate deafness interpreter service | 1

BASELINE CHARACTERISTICS:
Groups:
- Telephone-delivered Mindfulness: Participating Primary Caregivers and Care Partners receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
Arm/Group | Telephone-delivered Mindfulness
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  years
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers | 61 (9)
    Care Partners: number analyzed (Participants) | 28
    Care Partners | 53 (20)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers: Female | 26
    Primary Caregivers: Male | 3
    Care Partners: number analyzed (Participants) | 28
    Care Partners: Female | 19
    Care Partners: Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers: Hispanic or Latino | 1
    Primary Caregivers: Not Hispanic or Latino | 28
    Primary Caregivers: Unknown or Not Reported | 0
    Care Partners: number analyzed (Participants) | 28
    Care Partners: Hispanic or Latino | 0
    Care Partners: Not Hispanic or Latino | 28
    Care Partners: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers: American Indian or Alaska Native | 0
    Primary Caregivers: Asian | 0
    Primary Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Primary Caregivers: Black or African American | 29
    Primary Caregivers: White | 0
    Primary Caregivers: More than one race | 0
    Primary Caregivers: Unknown or Not Reported | 0
    Care Partners: number analyzed (Participants) | 28
    Care Partners: American Indian or Alaska Native | 0
    Care Partners: Asian | 0
    Care Partners: Native Hawaiian or Other Pacific Islander | 0
    Care Partners: Black or African American | 28
    Care Partners: White | 0
    Care Partners: More than one race | 0
    Care Partners: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Highest Education Level Completed [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers: High School or less | 2
    Primary Caregivers: Some College | 12
    Primary Caregivers: Bachelor's Degree | 10
    Primary Caregivers: Advanced Degree | 5
    Care Partners: number analyzed (Participants) | 28
    Care Partners: High School or less | 7
    Care Partners: Some College | 8
    Care Partners: Bachelor's Degree | 9
    Care Partners: Advanced Degree | 4
Number of Participants Working Outside the Home [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers | 15
    Care Partners: number analyzed (Participants) | 28
    Care Partners | 16
Annual Household Income [Count of Participants; unit: Participants] — Population: Data are reported separately for Primary Caregivers and Care Partners.
  Participants
    Primary Caregivers: number analyzed (Participants) | 29
    Primary Caregivers: Less than $20K per year | 9
    Primary Caregivers: $21-40K per year | 5
    Primary Caregivers: $41-60K per year | 6
    Primary Caregivers: $61-80K per year | 3
    Primary Caregivers: More than $80K per year | 3
    Primary Caregivers: Preferred Not to Answer | 3
    Care Partners: number analyzed (Participants) | 28
    Care Partners: Less than $20K per year | 4
    Care Partners: $21-40K per year | 10
    Care Partners: $41-60K per year | 4
    Care Partners: $61-80K per year | 3
    Care Partners: More than $80K per year | 4
    Care Partners: Preferred Not to Answer | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending at Least 6 Telephone Sessions
Description: The instructor will conduct a role call to take attendance at the beginning of each of the 8 class sessions and 1 retreat session. Eighty-five percent of participants who start the intervention will complete at least 6 out of 9 intervention sessions. Attendance used as a proxy to assess intervention acceptability.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Primary Caregivers: The primary caregivers providing regular daily care for a family member who has dementia receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
- Care Partners: A secondary informal caregiver who shares caregiving or helps make decisions regarding the person with dementia receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
- Total Population: Participating Primary Caregivers and Care Partners receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 29 | 28 | 57
Participants | 27 | 23 | 50

2. Primary Outcome: Percent of Dyads Who Endorse the Program
Description: The intervention will be acceptable to informal caregiving teams as evidenced by an 85 percent (95% Confidence Interval (CI): 72.5, 97.5) endorsement of the program in post-participation interviews. Calculated based on responses to open-ended questions regarding participants' experiences of the intervention. Examples of questions are: "how valuable or beneficial was the mindfulness training to you?" and "what challenges did you have with the training?" and "what did you expect from the training that you did not get?". Endorsement was considered positive if the expressions of value outweighed challenges (i.e., positive comments outweighed negative comments by dyad). Data reported as caregiving teams (dyads) in accordance with the protocol.
Time Frame: 8 weeks
Population: Of the 25 dyads completed, 1 Primary Caregiver and 1 Care Partner were unavailable to complete the interview thus eliminating 2 dyads and leaving 23 dyads for this evaluation.
Measure: Number; unit: percent of dyads
Arm/Group | Telephone-delivered Mindfulness
Number analyzed (Participants) | 46
percent of dyads | 100

3. Secondary Outcome: Change From Baseline in the Zarit Burden Interview Short Form (ZBI-12) Score
Description: The ZBI-12 is a 12-item (SF) version of the original 29-item questionnaire measures role strain and personal strain. Items are measured on a 5-point Likert scale (0=never to 4=nearly always). Scores range from 0-48 with lower scores representing less burden. Within group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: Two Care Partners are missing Baseline data due to an electronic glitch. One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 22 | 49
score on a scale | -2.5 [-4.5 to -0.5] | -3.6 [-6.6 to -0.5] | -2.9 [-4.5 to -1.3]

4. Secondary Outcome: Change From Baseline in the Family Satisfaction Scale (FSS) Score
Description: The FSS is a 10-item scale which uses a 5-point Likert scale (1=very dissatisfied to 5=extremely satisfied). Total scores range from 10-50 with higher scores representing more endorsement of family satisfaction. The FSS was administered at Baseline and Week 8. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: up to 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments and another Care Partner did not complete all of the measures.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 23 | 50
score on a scale | 2.78 [-0.70 to 6.25] | 4.30 [0.46 to 8.15] | 3.12 [0.75 to 5.50]

5. Secondary Outcome: Change From Baseline in Intolerance of Uncertainty Scale (IUS-12) Prospective Subscale Score
Description: The prospective anxiety subscale of the Intolerance of Uncertainty Scale (IUS-12) is a 7-item measure. The measure uses a 5-point Likert scale (1=not at all like me to 5=entirely like me). Scores range from 7-35, with lower scores reflecting more tolerance of uncertain situations. IUS-12 was administered at Baseline and at 8 weeks. Change scores are reported from paired t-tests for within-group assessments and from mixed effects models for the total population controlling for caregiving role, severity of dementia in the care recipient and dependencies in the data (individuals within families within cohorts).
Time Frame: up to 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a scale | -1.11 [-3.89 to 1.67] | -1.00 [-2.58 to 0.58] | -1.16 [-2.69 to 0.36]

6. Secondary Outcome: Change From Baseline in Intolerance of Uncertainty Scale (IUS-12) Inhibitory Subscale Score
Description: The inhibitory subscale of the Intolerance of Uncertainty Scale (IUS-12) is a 5-item measure. The measure uses a 5-point Likert scale (1=not at all like me to 5=entirely like me). Total scores range from 5-25, with lower scores reflecting more tolerance of uncertain situations. IUS-12 was administered at baseline and at 8 weeks. Within group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: up to 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Primary Caregivers: The primary caregivers provide regular daily care for a family member who has dementia.
- Care Partners: A secondary informal caregiver who shares caregiving or helps make decisions regarding the person with dementia.
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a scale | -0.81 [-2.22 to 0.59] | -1.17 [-2.47 to 0.14] | -0.97 [-1.87 to -0.09]

7. Secondary Outcome: Change From Baseline on PROMIS Meaning and Purpose-Short Form 6a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Meaning and Purpose-Short Form 6a is a 6-item scale that assesses a sense that life has purpose and there are good reasons for living, including hopefulness, optimism, goal-directedness, and feelings that one's life is worthy. It uses a 5-point Likert scale (1=strongly disagree to 5=strongly agree). Raw scores range from 6-30 with higher scores representing more endorsement of meaning and life. Raw scores are converted to T-scores based on population norms with a mean of 50 and standard deviation of 10. Therefore a score of 60 represents 1 standard deviation above the population average and indicates a high level of meaning and purpose. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: Data unavailable for one Care Partner who was unavailable at Week 8 and a Primary Caregiver who did not provide data at either Baseline or Week 8.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 26 | 24 | 50
T-score | 3.18 [0.52 to 5.85] | 2.23 [-0.84 to 5.29] | 2.7 [0.81 to 4.5]

8. Secondary Outcome: Change From Baseline on Cognitive and Affective Mindfulness Scale-Revised (CAMS-R)
Description: The CAMS-R is a 12-item scale measuring mindfulness by using language that is not representative of any particular meditation training or practice. It uses a 4-point Likert scale with responses ranging from 1 (Rarely/Not at all) to 4 (Almost always). Total scores range from 12-48. Higher scores indicate higher levels of mindfulness. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: The CAMS-R was added late and is unavailable at Baseline for the first 7 participants in the study (1st 4 Primary Caregivers, 1st 3 Care Partners). One Primary Caregiver did not complete the measure at Baseline or 8 weeks. One Care Partner who completed the intervention did not complete the measure at 8 weeks.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 22 | 21 | 43
units on a scale | 2.77 [0.22 to 5.32] | 2.04 [-0.22 to 4.31] | 2.5 [0.99 to 4.0]

9. Secondary Outcome: Change From Baseline on PROMIS Emotional Distress-Anxiety-Short Form 4a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety-Short Form 4a is a 4-item scale that assesses fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). It uses a 5-point Likert scale (1=never to 5=always). Raw scores range from 4-20 and are standardized to T-scores based on population averages (mean 50 and standard deviation 10). A score less than 55 is within normal limits. A score between 55-59.9 represents mild anxiety. A score greater than 60-69.9 represents moderate anxiety and a score of 70 or greater represents severe anxiety. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
T-score | -0.9 [-3.86 to 2.01] | 0.06 [-5.10 to 5.23] | 0.67 [-0.18 to 3.1]

10. Secondary Outcome: Change From Baseline on PROMIS Emotional Distress-Anger-Short Form 5a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anger-Short Form 5a item is a 5-item scale that assesses angry mood (irritability, frustration), negative social cognitions (interpersonal sensitivity, envy, disagreeableness), and efforts to control anger. It uses a 5-point Likert scale (1=never to 5=always). Raw scores range from 5-25 and are standardized to T-scores based on population averages (mean 50 and standard deviation 10). A score less than 55 is within normal limits. A score between 55-59.9 represents mild anger; 60-69.9 represents moderate anger and 70 or greater represents severe anger. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the study was unavailable to complete the post-intervention questionnaire.
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
T score | -0.79 [-3.89 to 2.30] | 2.21 [-2.11 to 6.54] | 0.67 [-1.8 to 3.1]

11. Secondary Outcome: Change From Baseline on PROMIS Global Physical Health
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Physical Health is a 2-item scale that assesses overall evaluation of one's physical health. It is based on the well-validated Rand measure, assessing general self-rated physical health, physical function, pain, and fatigue. It uses a 5-point Likert scale (1=poor to 5=excellent). Raw scores range from 2-10 and are standardized to T-scores with a population average of 50 and standard deviation of 10. Suggested cut points include 58 or higher = excellent; 50-57.9 = very good; 42-49.9 = good; 35-41.9 = fair, and less than 35 = poor. Change scores are reported from mixed effects models that utilize the entire population.
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: T score
Groups:
- Primary Caregivers: he primary caregivers providing regular daily care for a family member who has dementia receive mindfulness training in 8 weekly telephone sessions plus one retreat between weeks 5 and 6.
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
T score | -1.85 [-3.69 to -0.01] | -1.16 [-4.26 to 1.95] | -1.45 [-3.07 to 0.17]

12. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form is an 18-item measure consisting of 5 positive coping strategies (acceptance, positive refocusing, planning, positive reappraisal, putting into perspective) and 4 negative strategies (rumination, catastrophizing, self-blame, other-blame). Total scores range from 18-90 with higher scores representing more cognitive emotional regulation. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a scale | 1.48 [-0.82 to 3.78] | 0.88 [-2.68 to 4.42] | 1.29 [-0.59 to 3.16]

13. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Acceptance)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form acceptance subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater acceptance coping. Change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | 0.07 [-1.0 to 1.14] | -0.46 [-1.81 to 0.89] | -0.22 [-1.0 to 0.57]

14. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Positive Refocusing)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form positive refocusing subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater positive refocusing coping strategy. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | 0.15 [-0.84 to 1.13] | 1.08 [-0.52 to 2.68] | 0.55 [-0.30 to 1.4]

15. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Planning)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form planning subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater planning. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment. Another Care Partner declined to answer this question at Baseline.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 23 | 50
score on a subscale | 0.15 [-0.95 to 1.25] | -0.57 [-1.49 to 0.36] | -0.21 [-0.87 to 0.46]

16. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Positive Reappraisal)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form positive reappraisal subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater positive reappraisal. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | 0.07 [-0.75 to 0.90] | 0.25 [-0.53 to 1.03] | 0.25 [-0.29 to 0.78]

17. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Putting Into Perspective)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form putting into perspective subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater putting into perspective coping strategy. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | -0.41 [-1.41 to 0.59] | 0.67 [-0.68 to 2.01] | 0.23 [-0.53 to 1.0]

18. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Rumination)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form rumination subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater rumination. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | -1.0 [-1.87 to -0.13] | -0.04 [-0.94 to 0.85] | -0.49 [-1.1 to 0.1]

19. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Catastrophizing)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form catastrophizing subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater catastrophizing coping. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | -0.37 [-1.12 to 0.38] | -0.13 [-0.90 to 0.65] | -0.30 [-0.78 to 0.18]

20. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Self-Blame)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form self-blame subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater self-blame as a coping strategy. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving roles, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | -0.52 [-1.31 to 0.28] | 0.08 [-0.81 to 0.97] | -0.30 [-0.85 to 0.25]

21. Secondary Outcome: Change From Baseline on Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form (Other-Blame)
Description: Cognitive Emotional Regulation Questionnaire (CERQ)-Short Form other-blame subscale consisting of two questions. The subscale scores range from 2-10 with higher scores representing greater blaming others as a coping strategy. Change scores are reported from mixed effects models controlling for caregiving role, severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: score on a subscale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
score on a subscale | 0.11 [-0.52 to 0.74] | 0.21 [-0.58 to 1.00] | 0.14 [-0.31 to 0.60]

22. Secondary Outcome: Change From Baseline on PROMIS Emotional Support-Short Form 4a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support-Short Form 4a is a 4-item scale that assesses perceived feelings of being cared for and valued as a person and having confidant relationships. Item responses use a 5-point LIkert scale (1=never to 5=always). Raw scores range from 4-20. The PROMIS Emotional Support item is reported as a T score standardized to a population mean of 50 and standard deviation of 10 with higher scores reflecting more positive endorsement of emotional support. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessments and a Primary Caregiver completed only part of the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 26 | 24 | 50
T score | 0.48 [-2.29 to 3.21] | 1.39 [-2.43 to 5.21] | 0.89 [-1.22 to 3.0]

23. Secondary Outcome: Change From Baseline on PROMIS Informational Support-Short Form 4a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Informational Support-Short Form 4a is a 4-item scale that assesses perceived availability of helpful information or advice. Item responses use a 5-point LIkert scale (1=never to 5=always). Raw scores range from 4-20. The PROMIS Informational Support item is reported as a T score standardized to a population mean of 50 and standard deviation of 10 with higher scores reflecting more positive endorsement of informational support. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 26 | 24 | 50
T score | 2.72 [-0.83 to 6.27] | 2.05 [-1.83 to 5.93] | 2.65 [0.23 to 5.07]

24. Secondary Outcome: Change From Baseline on PROMIS Instrumental Support-Short Form 4a
Description: The PROMIS Instrumental Support-Short Form 4a is a 4-item scale that assesses perceived availability of assistance with material, cognitive or task performance. Item responses use a 5-point LIkert scale (1=never to 5=always). Raw scores range from 4-20. The PROMIS Instrumental Support item is reported as a T score standardized to a population mean of 50 and standard deviation of 10 with higher scores reflecting more positive endorsement of instrumental support. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 26 | 24 | 50
T score | 0.87 [-2.19 to 3.92] | 0.35 [-3.61 to 4.31] | 0.65 [-1.61 to 2.92]

25. Secondary Outcome: Change From Baseline on PROMIS General Self-Efficacy-Short Form 4a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) General Self-Efficacy-Short Form 4a is a 4-item scale that assesses confidence in ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. Items are measured on a 5-point Likert scale (1=I am not at all confident to 5=I am very confident). Raw scores range from 4-20. The PROMIS General Self-Efficacy item is reported as a T score standardized to a population mean of 50 and standard deviation of 10 with higher scores reflecting more positive endorsement of self-efficacy. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: T scores
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
T scores | 2.51 [-1.39 to 6.41] | 1.79 [-0.94 to 4.52] | 2.2 [-0.03 to 4.4]

26. Secondary Outcome: Change From Baseline in Mean NPI-Q Distress Scores
Description: The Neuropsychiatric Inventory (NPI-Q) Caregiver Distress subscale uses a 6-point scale with 12 items and scores ranging from 0-60. The NPI-Q measures the degree of distress associated with symptoms associated with dementia e.g., delusions, appetite change, and anxiety. Higher scores indicate more distress. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: Three Care Partners who provided no direct care did not complete this measure. One Care Partner who completed the intervention was unavailable to complete the post-intervention assessments. One Primary Caregiver did not complete the measure at Baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 26 | 21 | 47
units on a scale | -2.31 [-5.60 to 0.99] | -1.24 [-4.41 to 1.94] | -1.8 [-3.9 to 0.29]

27. Secondary Outcome: Change From Baseline on PROMIS Self-Efficacy for Managing Emotions-Short Form 4a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Emotions-Short Form 4a is a 4-item scale that assesses confidence to manage/control symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment and anger. Items are measured using a 5-point Likert scale (1=I am not at all confident to 5=I am very confident). Raw scores range from 4-20. The PROMIS Self-Efficacy for Managing Emotions item is reported as a T score standardized to a population mean of 50 and standard deviation of 10 with higher scores reflecting more positive endorsement of managing emotion. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 24 | 51
T score | 1.96 [-0.69 to 4.60] | -0.06 [-3.78 to 3.65] | 0.98 [-1.1 to 3.0]

28. Secondary Outcome: Change From Baseline in the Family Conflict Strategies for Care Subscale
Description: The FCS is a 12-item scale that measures the degree of conflict the family experiences about the seriousness of the care recipient's condition, concerns about the care recipient's safety, what the care recipient can do for him/herself, and whether a nursing home is indicated. The first subscale measures conflict around definitions of the illness and strategies for care (4 items). Items are measured on a 4-point Likert scale (1=no disagreement to 4=quite a bit of disagreement). The total scores range from 4-16 with lower scores representing less family conflict. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention did not complete the post-intervention assessments and another Care Partner completed only part of the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 23 | 50
score on a scale | -0.30 [-1.65 to 1.06] | -0.17 [-1.50 to 1.15] | -0.23 [-1.11 to 0.64]

29. Secondary Outcome: Change From Baseline in the Family Conflict Scale Attitudes and Actions Toward the Patient Subscale
Description: The FCS is a 12-item scale that measures the degree of conflict the family experiences about the seriousness of the care recipient's condition, concerns about the care recipient's safety, what the care recipient can do for him/herself, and whether a nursing home is indicated. The second subscale measures conflict around family members' attitudes and action toward the patient (4 items) Items are measured on a 4-point Likert scale (1=no disagreement to 4=quite a bit of disagreement). The total scores range from 4-16 with lower scores representing less family conflict. Within-group change scores are reported based on paired t-tests. Total change scores are reported from mixed effects models controlling for caregiving role, the severity of dementia in the care recipient, and dependencies in the data (individuals within families within cohorts).
Time Frame: Baseline, 8 weeks
Population: One Care Partner who completed the intervention was unavailable for the post-intervention assessments and another Care Partner completed only part of the post-intervention assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers | Care Partners | Total Population
Number analyzed (Participants) | 27 | 23 | 50
score on a scale | -0.30 [-1.95 to 1.35] | -0.43 [-1.94 to 1.07] | -0.34 [-1.35 to 0.68]

30. Secondary Outcome: Change From Baseline on Family Conflict Scale (FCS) Actions and Attitudes Toward the Caregiver Subscale
Description: The FCS is a 12-item scale that measures the degree of conflict the family experiences about the seriousness of the care recipient's condition, concerns about the care recipient's safety, what the care recipient can do for him/herself, and whether a nursing home is indicated. The third subscale measures conflict around family members' actions and attitudes around the caregiver (4 items). Items are measured on a 4-point Likert scale (1=no disagreement to 4=quite a bit of disagreement). The total scores range from 4-16 with lower scores representing less family conflict. This measure was requested from the primary caregiver only. Change scores are reported from mixed effects models controlling for the severity of dementia in the care recipient and dependencies in the data (individuals within cohorts).
Time Frame: Baseline, 8 weeks
Population: This subscale was administered only to the Primary Caregivers. Data was unavailable at follow-up for two Primary Caregivers who completed the intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Primary Caregivers
Number analyzed (Participants) | 25
score on a scale | -0.06 [-1.63 to 1.52]

ADVERSE EVENTS:
Time Frame: During the 8-week intervention period
Arm/Group | Primary Caregivers | Care Partners
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 2/29 | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Caregivers (N=29) | Care Partners (N=28)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional Distress (Psychiatric disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04058886/Prot_SAP_ICF_000.pdf